CLINICAL TRIAL: NCT00146406
Title: Integrated Multi-level Interventions to Improve Adolescent Health Through the Prevention of STD, Including HIV, and Teen Pregnancy
Brief Title: Multi-level Interventions for STD Prevention Among Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB terminated due to no continuation request.
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Health Research Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-4347; U30/CCU922283-01
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Chlamydia
Keywords: Adolescent Health; Sexually Transmitted Disease; Sexual Behavior
MeSH Terms: conditions — Chlamydia Infections; Sexually Transmitted Diseases; Sexual Behavior

INTERVENTIONS:
Behavioral: Project Connect

SUMMARY:
Sexually active adolescents between the ages of 10 and 19 are at extremely high risk for sexually transmitted diseases (STD), including HIV, and teen pregnancy.The overall goal of this research program is to develop, implement and evaluate integrated multi-level interventions to prevent STD, including HIV, and pregnancy among adolescents. The study includes 12 high schools and 19 of their feeder middle schools in the Los Angeles Unified School District and the surrounding communities. Interventions will be implemented among parents, health care providers, and in schools in an integrated fashion with the goal of improving social context factors related to health outcomes among adolescents. The evaluation phase will include in-school surveys with adolescents at all middle schools

DETAILED DESCRIPTION:
In the current study we plan to implement interventions at four social context levels, that is, with parents, providers or in other medical institutions, schools and community venues, to improve communication between adolescents and adults, facilitate increased access and utilization of health care services, and appropriate supervision of adolescents outside of school hours. As such the goals of the specific level interventions are as follows.

Among parents: (1) to enhance communication and relationship satisfaction; (2) increase parents participation in the healthcare of their adolescents; and (3) to enhance appropriate monitoring and supervision of adolescents.

Among school-based health care providers: (1) to increase access to and utilization of services by adolescents; and (2) to increase STD screening of adolescents.

In middle schools: (1) to increase access and utilization to supervised after-school activities, either at school or in the community; (2) to address quality and fidelity of health education curriculum provision and teacher training; (3) to increase parental participation in school-related activities.

In high schools: (1) to increase access and utilization to supervised after-school activities, either at school or in the community; (3) to address quality and fidelity of health education curriculum provision and teacher training; (4) to increase parental participation in school-related activities; (5) to increase awareness and utilization of school-based condom availability programs.

In community venues: (1) increase adolescents utilization of community-based clinical services; (2) to increase adolescent utilization of non-clinic-based screening; and (3) to increase utilization of community-based supervised activities for youth.

Activities will address these goals with the ultimate purpose of reducing adolescent risk for STDs, including HIV, and teen pregnancy through (1) increased age at first intercourse, (2) return to abstinence among sexually active adolescents, (3) decreased rates of unprotected sex among adolescents, (4) and increased screening and treatment of STD-infected adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Student at participating school

Exclusion Criteria:

* None

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36502 (Actual)
Dates: Start 2005-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Proportion of students who return to abstinence (measured yearly for 6 years)
Proportion of sexually active students who have unprotected intercourse (measured yearly for 6 years)
Proportion of sexually active students screened for chlamydia (measured yearly for 6 years)
Prevelance of chlamydia from Baseline to Year 6
Number of students who are sexually experienced (measured yearly for 6 years

SECONDARY OUTCOMES:
Parental monitoring (measured yearly for 6 years)
Parental communication (measured yearly for 6 years)
Supervision (measured yearly for 6 years)
Participation in after-school activities (measured yearly for 6 year)
Use of reproductive health care services (measured yearly for 6 years)

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Kerndt, M.D., Principal Investigator — Health Research Association
Locations (1):
- Health Research Association, Los Angeles, California, United States